CLINICAL TRIAL: NCT02722603
Title: Randomized, Double-blind, Double-dummy, Active Controlled, Multicentre, Non-inferiority Phase-III Study to Compare Gabapentin Liquid Formulation to Tramadol in Children Experiencing Moderate to Severe Chronic Neuropathic or Mixed Pain
Brief Title: Study to Compare Gabapentin to Tramadol in Children With Chronic Neuropathic or Mixed Pain
Acronym: GABA-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was early terminated due to insufficient recruitment
Sponsor: Pharmaceutical Research Management srl (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-004851-30
Record Dates: First submitted 2016-03-18; First posted 2016-03-30 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Gabapentin; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gabapentin / placebo tramadol (Experimental): gabapentin 75 mg/ml syrup / placebo tramadol, 3 times/day for 15 weeks.
  Interventions: Drug: gabapentin; Other: placebo tramadol
- tramadol / placebo gabapentin (Active Comparator): tramadol oral drops 100 mg/ml / placebo gabapentin, 3 times/day for 15 weeks.
  Interventions: Drug: tramadol; Other: placebo gabapentin

INTERVENTIONS:
Drug: gabapentin — 75 mg/ml gabapentin syrup
  Arms: gabapentin / placebo tramadol
Drug: tramadol — 100 mg/ml tramadol oral drops
  Arms: tramadol / placebo gabapentin
Other: placebo tramadol — placebo tramadol oral drops
  Arms: gabapentin / placebo tramadol
Other: placebo gabapentin — placebo gabapentin syrup
  Arms: tramadol / placebo gabapentin

SUMMARY:
This study evaluates the efficacy and safety of gabapentin relative to tramadol for the treatment of chronic, neuropathic or mixed pain in the paediatric population. Children from 3 months to less than 18 years of age experiencing moderate to severe chronic pain will receive either gabapentin or tramadol for 15 weeks. The difference in average pain scores between treatment arms at the end of the treatment period will be assessed.

DETAILED DESCRIPTION:
Gabapentin is indicated for the treatment of peripheral neuropathic pain in adults. In the absence of specific paediatric studies, it is not approved for the same condition in children.

The paediatric use of gabapentin is hampered by a) the lack of a suitable paediatric formulation, b) the significant variability of gabapentin pharmacokinetics profile and c) efficacy and safety data in this specific population.

The GABA-1 study is designed to demonstrate the efficacy of gabapentin oral solution relative to tramadol and to document the Pharmacokinetic and safety profile of gabapentin in this indication.

GABA-1 is a non-inferiority trial because gabapentin is expected to be equally effective but better tolerated than tramadol, thus providing a clinical benefit to affected children.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 3 months to less than 18 years at screening.
2. Informed consent by parent(s) and/or legal guardian according to each country legal requirement.
3. Assent by the patient, where applicable, according to each country legal requirement.
4. Subjects that meet the diagnostic criteria for neuropathic or mixed pain.
5. Subjects that present with chronic pain defined as the recurrent or continuous pain persisting more than 3 months. Duration of pain will be determined from the date of the first pain experienced.
6. Subjects that present with at least moderate pain as defined by average pain intensity of ≥4/10 as assessed during a 3-day screening period
7. Stable underlying disease condition and treatment.
8. In presence of malignant diseases, subjects in clinical remission and/or no expected changes in their therapeutic protocol during participation to the present study.

Exclusion Criteria:

1. Pain duration of more than 5 years.
2. Current use of gabapentin or tramadol.
3. History of failure to respond to adequate treatment by gabapentin or tramadol/opioids for neuropathic pain.
4. History of epileptic condition except febrile seizure disorder.
5. Subjects with sleeping apnoea syndrome of any origin or subjects with history of severe respiratory impairment.
6. Subjects with diagnosis of sickle cell disease.
7. Subjects that present significant cognitive impairment.
8. Subjects that present current, controlled or uncontrolled, co-morbid psychiatric diagnosis that can impair pain diagnosis and assessment such as severe depressive conditions or psychosis.
9. Subjects with history of suicidal ideation or behaviour.
10. History of substance abuse in particular opioids.
11. Subjects under prohibited concomitant medication
12. Subjects in need for corticosteroid oral treatment or corticosteroid infiltrations to treat pain caused by infiltration or compression of neural structures, e.g. peripheral nerves or spinal cord.
13. Subjects born prematurely at ≤ 36 weeks gestational age, if recruited during the first year of age.
14. Subjects with a body mass index (BMI) for age and gender of < 5th percentile or > 95th percentile.
15. Subjects with glomerular filtration rate < 90 mL/min/1.73 m2 (Schwarz equation).
16. Subjects with significant hepatic impairment or with Aspartate Transaminase (AST) or Alanine Transaminase (ALT) enzymes 3 times the upper limit of the age-specific reference range.
17. Subjects with known allergy, hypersensitivity or clinically significant intolerance to gabapentin or tramadol or any component found in the study drugs.
18. Subjects with fructose intolerance, diabetes, glucose-galactose malabsorption or lactase-isomaltase deficiency.
19. Subjects with clinically relevant abnormal ECG at the screening visit in the discretion of the Investigator/cardiologist.
20. Subjects participating in another clinical interventional trial.
21. Subjects scheduled for surgery or in recovery from surgery occurring within 3 months of baseline assessment.
22. Female subjects who are pregnant or currently lactating.
23. Subjects that failed screening or were previously enrolled in this study.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Pain score | an average of 16 weeks
  Pain score (0-10) measured at baseline (before starting the therapy) and at the end of the treatment in: patients aged 3-24 months using FLACC pain scale, patients aged 3-7 years using FPS-R scale, patients aged 8-17 years using NRS-11.
  The FLACC (the Faces, Legs, Arms, Cry and Consolability) scale is composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R (Faces Pain Scale - Revised - pts aged 3-7 years). Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11 (Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain.

SECONDARY OUTCOMES:
Percentage of responders to treatment | an average of 16 weeks
  Subjects with a pain intensity reduction of 30% from baseline or below or equal to 3/10, assessed by age-appropriate pain scale. FLACC (the Faces, Legs, Arms, Cry and Consolability) scale (pts aged 3-24-months) is composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R (Faces Pain Scale - Revised - pts aged 3-7 years). Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11 (Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain.
Daily pain intensity | an average of 3 weeks
  Daily pain intensity, assessed by age-appropriate scale (FLACC, FPS-R or NRS-11) during dose optimization.
  The FLACC (the Faces, Legs, Arms, Cry and Consolability) scale (pts aged 3-24-months) is composed by 5 categories. Each category is scored on the 0-2 scale, which results in a total score of 0-10, where 0=Relaxed and comfortable, 4-6=Moderate pain, 1-3=Mild discomfort, 7-10=Severe discomfort or pain or both.
  FPS-R (Faces Pain Scale - Revised - pts aged 3-7 years). Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
  NRS-11 (Numerical Rating Scale - pts aged 8-17 years): numerical rating scale where 0=no pain and 10=worst possible pain.
Observational assessment of pain | an average of 16 weeks
  Observational assessment of pain using the NRS-11 completed by parents and Investigator (or caregiver) at each visit.
  NRS-11: numerical rating scale where 0=no pain and 10=worst possible pain
Self-assessment of pain for children ≥8 years of age | an average of 16 weeks
  Self-assessment of pain for children ≥8 years of age using the FPS-R pain scale at each visit.
  FPS-R (Faces Pain Scale - Revised) Score is associated with face 0, 2, 4, 6, 8, or 10, where 0 = no pain and 10=very much pain.
Extent of pain | an average of 16 weeks
  number of painful areas using the pain charts at screening visit (V1), randomisation (v2) and EOS visit (V10). The pain charts are body maps (front and back) in which each body section is identified with a number.
Number of episodes of breakthrough pain | an average of 16 weeks
  Number of episodes of breakthrough pain (> 4/10 pain score and use of rescue medications) during treatment period.
Number of rescue interventions | an average of 15 weeks
  Number of rescue interventions required during treatment period
Number of pain-free days | an average of 15 weeks
  Number of pain-free (< 4/10 average pain score without the use of rescue medications) days during treatment period
Number of participant dropouts | up to 21 weeks
  Number of participant dropouts due to lack of efficacy
The total cumulative weight normalized dose of each rescue drug | up to 21 weeks
  The total cumulative weight normalized dose of each rescue drug
Total Summary Score from PedsQL™ scale | an average of 15 weeks
  Total score obtained using the PedsQL 4.0 Generic Core Scales (by parent, patient aged 3-17years) and PedsQL Infants Scales (by parent of pts aged 3-24months) at randomisation (V2) and at EOS (V10). The total score is a measure of Health Related Quality of life (HRQoL). Higher scores indicate better HRQOL.
  PedsQL 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL Infant Scales is composed by 5 multidim. scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always)
Physical Health Summary Score from PedsQL™ scale | an average of 15 weeks
  Physical Health Score obtained using the PedsQL™ 4.0 Generic Core Scales (by parent, patient aged 3-17 years) and PedsQL™ Infant Scales (by parent, aged 3-24 months) at randomisation (V2) and at EOS (V10).
  PedsQL™ 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL™ Infant Scales is composed by 5 multidimensional scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
Psychosocial Health Summary Score from PedsQL™ scale | an average of 15 weeks
  Psychosocial Health Score obtained using the PedsQL™ 4.0 Generic Core Scales (by parent, patient aged 3-17 years) and PedsQL™ Infant Scales (by parent, aged 3-24 months) at randomisation (V2) and at EOS (V10).
  PedsQL™ 4.0 Generic Core Scales is composed by 4 multidimensional scales (Physical Funct, Emotional Funct, Social Funct, School Funct) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). Scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
  PedsQL™ Infant Scales is composed by 5 multidimensional scales (Physical Functioning, Physical Symptoms, Emotional Functioning, Social Functioning, Cognitive Functioning) and 3 summary scores (Total Scale Score, Physical Health Summary Score, Psychosocial Health Summary Score). The scoring is based on a 5-point Likert scale from 0 (Never) to 4 (Almost always).
Acceptability of treatment | at week 16
  Acceptability of treatment (Five-Point Facial Hedonic scale) at EOS visit (V10).
  Each face in the scale is related to a score (1=unpleasant; 2=not sure; 3=pleasant).
Global satisfaction with treatment | at week 15
  Global satisfaction with treatment (NRS-11, by parent, patient) at EOS visit (V10).
  The satisfaction is measeured by the numerical rating scale NRS-11 where 0=not satisfied and 10=fully satisfied
Clinical Global Impression of Severity of the subject's condition | an average of 15 weeks
  Clinical Global Impression of Severity (CGI-S) for Neuropathic or Mixed Pain Overall Severity Prior to Study Treatment (at randomization - V2) assessed by Investigator.
  Investigators will rate their impression of the severity of the subject's condition. Scoring: Normal: no signs of pain, Borderline painful, Mildly painful, Moderately painful, Markedly painful,Severely painful, Among the most extremely painful patients.
Clinical Global Impression of Improvement for pain | an average of 15 weeks
  Clinical Global Impression of Improvement (CGI-I) for Neuropathic or Mixed Pain Overall at V6 and EOS visit (V10) assessed by Investigator.
  Investigators will rate their impression of any change of the subject's overall condition of neuropathic or mixed pain since randomization in the study. Scoring are: Very much improved since the initiation of treatment; Much improved; Minimally improved; No change from baseline (the initiation of treatment); Minimally worse; Much worse; Very much worse since the initiation of treatment.
Patient/parent Global Impression of Change | an average of 12 weeks
  Patient/parent Global Impression of Change (PGIC; by parent, patient) at V6 and at EOS visit (V10).
  Patient/parent will rate their impression of any change of the subject's overall condition of neuropathic or mixed pain since randomization in the study. Scoring are: Very much improved since the initiation of treatment; Much improved; Minimally improved; No change from baseline (the initiation of treatment); Minimally worse; Much worse; Very much worse since the initiation of treatment.
CL/F | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameters for gabapentin and tramadol: assessment of apparent clearance (CL/F) and of its variability and precision. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Vd/F | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameter for gabapentin and tramadol: assessment of apparent volume of distribution (Vd/F) and of its variability and precision. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
ka | at week 3 or at week 4 or at week 16
  Primary pharmacokinetic parameter for gabapentin and tramadol: assessment of absorption rate constant (Ka) and of its precision and variability. In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
AUC | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin and tramadol: assessment of Area under the Concentration curve (AUC). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Cmax | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin and tramadol: assessment of peak plasma concentration (Cmax). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Tmax | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin and tramadol: assessment of time at which the Cmax is observed (Tmax). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Css | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin and tramadol: assessment of steady state Concentrations (Css). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Cmin | at week 3 or at week 4 or at week 16
  Secondary pharmacokinetic parameter for gabapentin and tramadol: assessment of minimum concentration (Cmin). In total, 4 samples will be collected, 1 before dosing and again at 3 different time windows post-dosing (0 - 2 h; 2 - 4 h and 4 - 6 h)
Systemic exposure to investigational products during maintenance period | an average of 12 weeks
  Systemic exposure to investigational products during maintenance period, as assessed by predicted steady-state concentrations.
Incidence of Adverse Events at all visits | up to 21 weeks
  Incidence of Adverse Events at all visits
Percentage of subjects discontinuing the trial due to treatment-emergent adverse events. | up to 21 weeks
  Percentage of subjects discontinuing the trial due to treatment-emergent adverse events.
Aggressive behaviour in children aged >6 years | an average of 15 weeks
  Aggressive behaviour in children aged >6 years using the Retrospective-Modified Overt Aggression Scale (R-MOAS) at V2, V6 and EOS visit (V10).
  The scale includes 4 domains (Verbal Incidents, Incidents Toward Other People, Incidents Involving Property, Incidents Directed Toward Self) each one describing different behaviours.
  Parents rate the frequency of 16 aggressive behaviors (referred to the past week) in the 4 areas. Numeric weighting amplifies the seriousness of more harmful behaviors in the total score. Higher score indicating more aggressive behavior.
Suicidal ideation/behaviour in subjects aged 6 years and older | an average of 16 weeks
  Suicidal ideation/behaviour in subjects aged ≥ 6 years using the Columbia - Suicide Severity Rating Scale (C-SSRS) before IMP (screening V1), V6, EOS visit (V10) and end of taper visit (V11). The C-SSRS is divided into 2 sections: Suicidal Ideation and Suicidal Behaviour containing each one 5 "yes" or "no" questions.
  Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the CSSRS) present at the assessment. A score of 0 is assigned if no ideation is present.
  Composite endpoints are defined below:
  Suicidal ideation: A "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5).
  Suicidal behavior: A "yes" answer at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10).
  Suicidal ideation or behavior: A "yes" answer at any time during treatment to any one of the ten suicidal ideation and behavior questions (Categories 1-10)
Assessment of blinding | at week 16
  Assessment of blinding: guess of the subject's treatment group (by Investigator, parents and subject if at adequate maturity level) at V10.

CONTACTS AND LOCATIONS:
Overall Officials: Florentia Kaguelidou, Principal Investigator — Center Clin Investig INSERM CIC 1426 H. R Debré APH de Paris
Locations (2):
- Universitaets klinikum Erlangen, Erlangen, Germany
- Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam, Netherlands

REFERENCES:
- [Background] Finnerup NB, Sindrup SH, Jensen TS. Recent advances in pharmacological treatment of neuropathic pain. F1000 Med Rep. 2010 Jul 14;2:52. doi: 10.3410/M2-52. PMID 21170362
- [Background] Mellegers MA, Furlan AD, Mailis A. Gabapentin for neuropathic pain: systematic review of controlled and uncontrolled literature. Clin J Pain. 2001 Dec;17(4):284-95. doi: 10.1097/00002508-200112000-00002. PMID 11783808
- [Derived] Kaguelidou F, Le Roux E, Mangiarini L, Lundin R, de Leeuw TG, Della Pasqua O, Felisi M, Bonifazi D, Tibboel D, Ceci A, de Wildt SN, Alberti C; GAPP consortium. Non-inferiority double-blind randomised controlled trial comparing gabapentin versus tramadol for the treatment of chronic neuropathic or mixed pain in children and adolescents: the GABA-1 trial-a study protocol. BMJ Open. 2019 Feb 20;9(2):e023296. doi: 10.1136/bmjopen-2018-023296. PMID 30787078